CLINICAL TRIAL: NCT05729191
Title: Evaluation of the Acceptance of the Anti-COVID-19 Vaccine Offer and of the Knowledge and Attitudes Towards the Vaccination Among Pregnant Women Through a Validation Study at the Fondazione Policlinico Universitario A IRCCS Twins (FPG).
Brief Title: Evaluation of the Acceptance of the Anti-COVID-19 Vaccine Offer Among Pregnant Women
Status: Completed | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Bruno Stefania, Medical Doctor Specialized In Hygiene and Preventive Medicine, Researcher, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 4557
Record Dates: First submitted 2023-02-14; First posted 2023-02-15 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Pregnant Women; COVID 19 Vaccine; Vaccination Hesitancy
MeSH Terms: conditions — Vaccination Hesitancy

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: Anti Covid 19 vaccination campaign for pregnat women — Assessment of vaccine hesitancy and Covid-19 disease knowledge

SUMMARY:
The SARS-CoV-2 pandemic still represents a global health, social and economic emergency. In Italy, since the beginning of the pandemic, a total of 4,709,753 cases and 131,461 deaths have been recorded.

The vaccination campaign against COVID-19, launched on 27 December 2020, has made it possible in Italy to achieve complete vaccination coverage (two doses) of 80.6% of the population aged > 12 years. The latest data on the impact of vaccination in preventing new infections, hospitalizations and deaths report a strong reduction in the risk of SARS-CoV-2 infection in fully vaccinated people compared to unvaccinated people (78% for diagnosis, 92% for hospitalization, 95% for ICU admissions and 94% for deaths); most of the cases notified in the last 30 days in Italy have been diagnosed in unvaccinated people2.

Evidence on the immunogenicity and safety of anti-SARS-CoV-2 vaccination in pregnant women, although not deriving from clinical trials, is growing, even if not yet conclusive. On the efficacy of mRNA vaccines in pregnancy, a retrospective Israeli cohort study reported a significantly lower risk of contracting SARS-CoV-2 infection compared to unvaccinated women. Furthermore, a greater maternal and perinatal morbidity from COVID-19, also associated with the circulation of the Delta variant, has been highlighted by the recent analyzes of the English data, updated to 11 July 2021.

The Istituto Superiore di Sanità, in the light of the growing evidence on the safety of vaccination during pregnancy for both the fetus and the mother, the new evidence relating to the greater morbidity associated with the Delta variant, the growing circulation of the same variant and the significant lowering of median age at infection in Italy, recommends extending the vaccine offer, with mRNA vaccines, to all pregnant women in the second and third trimester.

Objectives of the study: Evaluate the quality in terms of reception of the anti-COVID-19 vaccine offer, the knowledge and attitudes towards the aforementioned vaccination by pregnant women who join the Vaccination Open Day and who access the FPG Covid Vaccination Center for this vaccination.

Primary endpoint: Measuring acceptance of the anti-COVID-19 vaccine offer and knowledge about vaccination, by means of a questionnaire to be administered after vaccination.

DETAILED DESCRIPTION:
Background Evidence on the immunogenicity and safety of anti-SARS-CoV-2 vaccination in pregnant women, although not deriving from clinical trials, is growing, even if not yet conclusive. On the efficacy of mRNA vaccines in pregnancy, a retrospective Israeli cohort study reported a significantly lower risk of contracting SARS-CoV-2 infection compared to unvaccinated women. Furthermore, a greater maternal and perinatal morbidity from COVID-19, also associated with the circulation of the Delta variant, has been highlighted by the recent analyzes of the English data, updated to 11 July 2021.

The Istituto Superiore di Sanità, in the light of the growing evidence on the safety of vaccination during pregnancy for both the fetus and the mother, the new evidence relating to the greater morbidity associated with the Delta variant, the growing circulation of the same variant and the significant lowering of median age at infection in Italy, recommends the extension of the vaccination offer, with mRNA vaccines, to all pregnant women in the second and third trimester. Although vaccination can be considered throughout pregnancy, a benefit-risk assessment with a physician is recommended for women wishing to be vaccinated in the first trimester, as there is still little evidence relating to this gestational age. Finally, the same document identifies the priority target for vaccination in pregnancy:

* women at increased risk of contracting SARS-CoV-2 infection (e.g. health professionals, caregivers)
* and/or at greater risk of developing a serious disease from COVID-19 (women with risk factors: age >30 years, BMI >30, comorbidities, citizenship of countries with high migratory pressure), with possible repercussions also on the outcomes fetus/ neonates.

Project phases

The study includes six implementation phases:

1. Preliminary stage

   * Establishment of the working group for sharing and planning activities.
   * Analysis of literature data to define the context, the target population and the current status of anti-SARS-CoV-2 vaccination in pregnant women.
2. Start up with creation, on the day of the Open Day, an anti-COVID-19 vaccine awareness event for those enrolled in the active childbirth preparation course at the A. Gemelli IRCCS Polyclinic Foundation (from now on referred to as FPG), including:

   * Training interventions and testimonials on the anti-COVID-19 vaccination and the impact of the infection on pregnant women.
   * Preparation of a questionnaire relating to the approval of the vaccination offer on the occasion of the vaccination Open Day and to the knowledge in the field of vaccination to be submitted after the administration of the vaccination, during the observation period.
   * Creation of informative material (poster).
3. Vaccination administration, scheduled for 25 October 2021. The vaccination will be administered by the nursing staff of the FPG and by doctors in specialist training in hygiene and preventive medicine and doctors of the UOC Hospital Hygiene, after collection of informed consent.
4. Administration of the questionnaire after vaccination.
5. Possible expansion of the sample of pregnant women at the FPG Covid Vaccination Center.
6. Analysis of the results achieved - Calculation of study endpoints and disclosure of the same.

Human and financial resources

The human resources used to carry out the activities listed above will be represented by:

* Doctors in specialist training in Hygiene and Preventive Medicine (as part of the professionalizing activity of the Hospital Hygiene Unit),
* FPG nursing staff,
* Medical directors of the UOC of Hospital Hygiene and of the UOC of Obstetrics and Gynecology No additional costs will be required from the FPG for the conduct and management of the study as the vaccines will be offered free of charge by the Region and ASL Roma 1 (National Health System).

OBJECTIVES AND ENDPOINTS

Primary objective: Evaluate the quality in terms of reception of the anti-COVID-19 vaccine offer by pregnant women who join the vaccination Open Day and their knowledge and attitudes towards the aforementioned vaccination.

Primary endpoint: Measure the liking of the anti-COVID-19 vaccine offer and knowledge about vaccination, by means of a questionnaire to be administered after vaccination.

STUDY DESIGN AND PLANNING

Study design Single center observational prospective exploratory.

Setting "A. Gemelli IRCSS.

Study population The population included in the study is represented by pregnant women who will join the vaccination offer, recruited from those enrolled in the childbirth preparation course, organized by the UOC of Obstetrics and Obstetric Pathology of the FPG and/or belonging to the Covid FPG Vaccination Center.

Duration of the study One year: the vaccination Open Day will be held on October 25; the questionnaire will be administered on the same date; if it is necessary to expand the sample, the duration will also be extended to the FPG Covid Vaccination Center. Subsequently, the data processing will be carried out.

Sample size Given the exploratory nature of the study, a formal calculation of sample size is not required. The sample is of opportunity. On the basis of the number of pregnant patients attending the course of preparation for childbirth, organized by the UOC of Gynecology and Obstetrics, at the FPG, the enrollment of about 100 subjects is expected.

Data collection and sources The results of the completed questionnaires will be digitized in a special Excel electronic database by doctors belonging to the Hospital Hygiene Unit. This database will be used for the analysis of data relating to the questionnaires. The data will be anonymised and the results will be presented in aggregate form.

Data management and statistical analysis As this is an exploratory study, the data will be analyzed exclusively using descriptive statistics indices.

In detail, the qualitative variables will be represented as absolute frequencies and percentages. The quantitative variables will be evaluated through the Shapiro-Wilk test, to verify the normality of the distribution. In case of normally distributed data, they will be expressed as mean and standard deviation (SD); otherwise, by median and interquartile range (IQR).

The analyzes will be conducted using STATA software version 16.

Data processing and protection The study will be conducted in accordance with Good Clinical Practice, the Declaration of Helsinki and all applicable legislation in the field of this matter. The data will be processed anonymously and presented in an aggregated manner, according to privacy protection criteria already in place at FPG.

Informed consent The informed consent form for participation in the study and the use of data relating to treatment for research needs will be given to all those who agree to complete the questionnaire following the vaccination on the Open Day of 25 October 2021. as required by this Ethics Committee.

ELIGIBILITY:
Inclusion Criteria:

* The population included in the study is represented by pregnant women who will join the vaccination offer, recruited from those enrolled in the childbirth preparation course, organized by the UOC of Obstetrics and Obstetric Pathology of the FPG and/or belonging to the Covid FPG Vaccination Center.

Exclusion Criteria:

- Pregnant women under 18 years old

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant women
Study Population: The population included in the study is represented by pregnant women who will join the vaccination offer, recruited from those enrolled in the childbirth preparation course, organized by the UOC of Obstetrics and Obstetric Pathology of the FPG and/or belonging to the Covid FPG Vaccination Center.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-10-25 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-03-30 (Actual)

PRIMARY OUTCOMES:
Compliance and knowledge | 2021-2022
  Measure the acceptance of the anti-COVID-19 vaccine offer and knowledge about vaccination, by means of a questionnaire to be administered after vaccination.

CONTACTS AND LOCATIONS:
Overall Officials: Stefania Bruno, edicine, Principal Investigator — Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Locations (1):
- Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Roma, Italy

IPD SHARING:
Plan to Share IPD: No
aggregated data could be published with a scientific paper